CLINICAL TRIAL: NCT01384305
Title: Establish a "Taiwan Rare Disorder Tissue Bank", to Collect and Repost Biological Samples and Disease Information From Patients With Rare Disorders
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: China Medical University Hospital (Other)
Responsible Party: China Medical University Hospital, China Medical University Hospital
Other Study IDs: DMR98-IRB-255-3
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Rare Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Even though rare disorders usually have limited case numbers, they have induced huge impacts on patients and their families, and has heavily burdened on our society and healthcare system as well. Therefore, it is essential to detect the occurrence of disorders and thus take appropriate measures as early as possible. The preventive goal is based on comprehensive understanding on rare disorders, available diagnostic and therapeutic approaches. However, studies related to rare disorders are often impeded by limited sample sizes and infrequent exchange of research materials among institutes. After referring to foreign experiences, the investigators have noticed that a non-profit tissue bank which can reposit biological samples and thus provide researchers access to samples, may be a solution. Through sharing this public asset, the investigators believe not only quantity and quality of rare disorder studies will be improved, the collaboration between various research institutes can also be strengthened afterwards. Most important of all, those achievements can ultimately benefit patients, families and the whole society.

DETAILED DESCRIPTION:
Investigation Plan

1. Study Period：From 2009 to 2013
2. Study Population：Patients with rare disorders.
3. Planned Number of Subjects： 300~500 Subjects will be included in CMU.
4. Inclusive Criteria：A patient who is clinically diagnosed as one of rare disorders notified by Department of Health or our organization. Or a patient who is diagnosed as a probable rare disorder case by physicians.
5. Exclusive Criteria：Patients whose physical or mental status is not suitable by the judgment of health professionals. Or a patient who is <20 years old or interdictory, yet without getting the permission from his/her legal representatives.
6. Study Site： Mainly in OPD that related to rare disorders.
7. Study Materials：Blood (for plasma, DNA and cell line), a questionnaire and a chart review form. Tissue samples are acceptable as well.
8. Application of collected materials：Samples and information will be restored in appropriate manner, and researchers will be encouraged to apply them for biological studies in the field of rare disorders thereafter.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is clinically diagnosed as one of rare disorders notified by Department of Health or our organization. Or a patient who is diagnosed as a probable rare disorder case by physicians.

Exclusion Criteria:

* Patients whose physical or mental status is not suitable by the judgment of health professionals. Or a patient who is < 20 years old or interdictory, yet without getting the permission from his/her legal representatives.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rare disorders.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-12